CLINICAL TRIAL: NCT03346746
Title: Utilizing GI: Exploring an Optimum Glycaemic Profile for Cognitive Function Across the Day in Healthy Individuals
Brief Title: Utilizing GI: Exploring an Optimum Glycaemic Profile for Cognitive Function Across the Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Grout (Other)
Responsible Party: Sponsor-Investigator, Matthew Grout, Doctoral Researcher, University of Reading
Organization: University of Reading (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-206-DL
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Cognitive Performance; Glucose, Low Blood; Glucose, High Blood; Mood
Keywords: cognition; glycaemic; mood; diet

STUDY DESIGN:
Intervention Model Description: All participants took part in both conditions.
Who Masked: Participant
Masking Description: Participants were not told what diet they were consuming each day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low GI diet (Experimental): This diet contained three Low GI meals. This was the Low Glycaemic Diet intervention.
  Interventions: Dietary Supplement: Low Glycaemic Diet
- High GI diet (Experimental): This diet contained three meals, all with a high GI value. This was the High Glycaemic Diet intervention.
  Interventions: Dietary Supplement: High Glycaemic Diet

INTERVENTIONS:
Dietary Supplement: Low Glycaemic Diet — This intervention was a diet that provided participants with three meals with a low GI value. These meals were breakfast (9am), lunch (midday) and a snack (3pm).
  Arms: Low GI diet
Dietary Supplement: High Glycaemic Diet — This intervention was a diet that provided participants with three meals with a high GI value. These meals were breakfast (9am), lunch (midday) and a snack (3pm).
  Arms: High GI diet

SUMMARY:
This study provides participants with two diets that vary in their glycaemic index values (low vs. high), whilst also measuring cognitive performance and mood.

DETAILED DESCRIPTION:
Therefore, the current study introduces cognitive testing into study procedures. Participants will consume the favourable and unfavourable conditions (each containing three meals) on separate days following a crossover, randomised, couterbalanced design. The primary dependent variable is cognitive function, whilst secondary measures include glucose and mood. It is hypothesised that the favourable meal profile will be associated with cognitive and physiological benefits relative to the unfavourable meal profile.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 25 years of age
* Willing to participate in the entire study (signed informed consent required)
* Male or female (not pregnant)

Exclusion Criteria:

* Suffer from diabetes
* Are anaemic
* Smoker
* Have any food intolerances or allergies
* History of alcohol or drug misuse
* Diagnosed with any of the following;

  * High blood cholesterol
  * High blood pressure
  * Thyroid disorder
  * Heart problems, stroke or any vascular disease in the past 12 months
  * Inflammatory diseases such as rheumatoid arthritis
  * Bone related conditions, such as osteoporosis
  * Renal, gastrointestinal, respiratory, liver disease or cancer
* You are presently taking part in another clinical trial or research study
* You are an elite athlete (very high intensity training more than 3 times a week)
* You are currently on a specific diet, and are unwilling to cease during the testing period
* You are intending to regularly use medication which affects gastrointestinal motility

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance between time points assessed | This was tested 9 times a day, with two days, giving a total of 18 times. Each battery of four tasks lasted approximately 15 minutes
  A participants performance over four cognitive tasks

SECONDARY OUTCOMES:
Glycaemic profile | This was measured 23 times a day, for two days, giving a total of 46 times
  Glucose concentration levels
Mood (alertness, anxiety and contentment) using the Bond-Lader (1974) Visual Analogue Scale | This takes approximately 5 minutes to complete. Participants were tested six times a day. There were two test days. Giving a total of 12 times, or approximately 60 minutes of mood scale completion.
  This was comprised of three mood sub-factors; alertness, anxiety, contentment. The VAS provides participants with 16 lines (100mm in length). At each end of every line are two words opposite in meaning, for example 'alert' and 'drowsy'. A participant marks each line closer to the word they feel at that current time. The minimum score is 0 and the maximum is 100, measured in millimetres.
Sleepiness | This takes approximately 30 seconds to complete. Participants were tested six times a day. There were two test days. Giving a total of 12 times, or approximately 6 minutes overall.
  This was measured on a custom Visual Analogue Scale. Participants were presented with a 100mm line. At one end the word 'sleepy' appeared, and at the other end 'not sleepy' was present. Participants indicated how sleepy they felt by marking the line closer to the word they currently felt. Scores fell between 0 and 100.
Hunger | This takes approximately 30 seconds to complete. Participants were tested six times a day. There were two test days. Giving a total of 12 times, or approximately 6 minutes overall.
  This was measured on a custom Visual Analogue Scale. Participants were presented with a 100mm line. At one end the word 'hungry' appeared, and at the other end 'not hungry' was present. Participants indicated how hungry they felt by marking the line closer to the word they currently felt. Scores fell between 0 and 100.
Fullness | This takes approximately 30 seconds to complete. Participants were tested six times a day. There were two test days. Giving a total of 12 times, or approximately 6 minutes overall.
  This was measured on a custom Visual Analogue Scale. Participants were presented with a 100mm line. At one end the word 'full' appeared, and at the other end 'not full' was present. Participants indicated how full they felt by marking the line closer to the word they currently felt. Scores fell between 0 and 100.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Lamport, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No